CLINICAL TRIAL: NCT02024672
Title: Ultrasound Surveillance of IUDs Placed Immediately Postpartum
Brief Title: Monitoring With Ultrasound Imaging of Intrauterine Device (IUD) Position Placed Immediately After Giving Birth
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Other Study IDs: GCO 13-1557
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Contraception; Postpartum
Keywords: Intrauterine devices; IUDs; postpartum; contraception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Immediate postpartum placement of IUD: Women who plan to have an IUD placed at the time of cesarean section or vaginal delivery, or women who have had an IUD placed at the time of cesarean section or vaginal delivery.
  Interventions: Other: Immediate postpartum placement of IUD

INTERVENTIONS:
Other: Immediate postpartum placement of IUD — pelvic exam, transvaginal ultrasound (3 during the course of the study), bleeding and symptom diary

SUMMARY:
Intrauterine devices (IUDs) are one of the most effective reversible forms of contraception, and are a good option in the postpartum period for women to avoid a rapid repeat pregnancy. IUDs can be placed immediately postpartum, after delivery of the placenta by either vaginal or cesarean birth. This practice has been shown to be safe, and is recommended by the American College of Obstetricians & Gynecologists, the World Health Organization and the U.S. Center for Disease Control. Immediate postpartum IUD placement has the advantage of providing contraception at a time that the woman is already accessing medical care, avoiding potential loss to follow up or risk of unintended pregnancy. Additionally, women who have anesthesia for delivery have reduced pain at the time of IUD placement compared to having the IUD placed at the postpartum follow up appointment. Immediate postpartum IUD placement is a relatively new practice in the US and little is known about the expected appearance of IUDs inside the uterus taken with an ultrasound when they have been placed at the time of delivery. It is less likely that IUD strings will be visible at the cervix after immediate postpartum IUD placement due to subsequent uterine involution, which makes it important to monitor correct positioning of the IUD via ultrasound. This study will document normal changes in the positioning of the IUD visualized via ultrasound, and determine if a correlation exists between IUD position and risk of expulsion. Ultrasound surveillance to document IUD position and distance from the fundus, will be performed at 6 weeks, 3 months and 12 months after placement. Symptoms of menstrual bleeding and pain will also be recorded in order to determine if they are correlated with IUD position.

DETAILED DESCRIPTION:
The goal of this study is to document the expected ultrasound appearance of intrauterine devices (IUDs) placed immediately postpartum. This practice has been shown to be safe and effective, but little is known about long-term follow up for IUDs placed in this setting. Because IUD strings will not be visualized for many patients after immediate postpartum IUD placement, sonographic imaging will likely be required for the majority of patients to determine expulsion. However, the ultrasound appearance of these IUDs, placed immediately after birth and before uterine involution, may be different than those IUDs placed outside of the postpartum period. To our knowledge no other study has documented expected ultrasound appearance of IUDs placed in the immediate postpartum period.

The specific aims of this study are to: 1. document normal appearance of IUDs on ultrasound after immediate postpartum placement; 2. document if this appearance changes over time; and 3. determine if location on ultrasound is associated with side effects or expulsion.

Study design This is a prospective, observational study. All patients who have an IUD (either copper or levonorgestrel) placed immediately postpartum (within 10 minutes of delivery of placenta) after either Cesarean or vaginal delivery at Mount Sinai Medical Center and at Elmhurst Hospital Center will be eligible to participate in the study.

Study visits will include a speculum exam for IUD string check at 6 weeks, and ultrasounds to evaluate IUD position at the following time points: 6-10 weeks following placement, 3 months following placement (with inclusion up to 6 months), and 12 months following placement (with inclusion up to 15 months).

The ultrasound will document the following: size and position of uterus, IUD-Myometrium distance, IUD-endometrium distance, IUD-fundus distance and position of IUD. When participants present for the scheduled ultrasound visits, they will be asked to return with the completed symptom diary as well, to assess bleeding and pain.

Study Endpoints IUD expulsion, removal, or completion of the 12-15 month follow up visit will be the study endpoints. The participant will be withdrawn from the study if IUD expulsion occurs, or if she requests IUD removal for any reason. Participants will also be able to withdraw from the study at any time if they no longer wish to participate, but they may keep their IUD in place if desired.

Study procedures At the routine 6 week postpartum visit for all patients, pelvic and speculum exam will be performed as per normal clinical routine, and visualization of IUD strings at the cervical os will be documented. If IUD strings are not visualized, an ultrasound will be performed by the clinical provider to confirm presence or absence of IUD within the uterus.

A formal ultrasound to evaluate IUD position will be scheduled in the FPA gynecologic ultrasound unit or in the Gynecology clinic at EHC at the following time points: 6-10 weeks following placement, 3 months following placement (with inclusion up to 6 months), and 12 months following placement (with inclusion up to 15 months). The formal ultrasound will document the following: size and position of uterus, endometrial stripe (EMS) thickness, IUD-Myometrium distance, IUD-endometrium distance, IUD-fundus distance and position of IUD.

Immediate postpartum placement of IUDs is a relatively new clinical practice in the United States; as such there is no recommended or "standard" follow up protocol in this situation. For IUDs placed outside of the postpartum period, the standard follow up is a string check (speculum exam to confirm presence of strings at cervical os) 2-6 weeks after IUD placement. If strings are not visible, or if the patient experiences symptoms concerning for expulsion, a transvaginal ultrasound will be performed. Once correct placement is confirmed by ultrasound, patients without visible strings generally have ultrasounds yearly to confirm placement. Based on this standard practice, patients with visible strings will have the ultrasound only for research purposes. Additionally, the three month ultrasound will be only for research purposes, even in those without visible strings.

When participants present for the scheduled ultrasound visits, they will be asked to return with the completed symptom diary as well.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years of age
* English or Spanish speaking
* Desire postpartum IUD placement, either copper IUD or levonorgestrel IUD

Exclusion Criteria:

* Contraindications for IUD use (CDC MEDICAL Eligibility Criteria category 3 or 4 for specific IUD)
* Positive Chlamydia or gonorrhea cervical cultures in past 3 months
* Immediate postpartum hemorrhage
* Premature rupture of membranes (PROM) >12h or diagnosis of endometritis

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from the group of women receiving prenatal care at Mount Sinai Hospital in New York City and Elmhurst Hospital in Queens. Patients who express an interest in an IUD for contraception after delivery will be given information about immediate postpartum IUDs and the study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2013-12; Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
IUD-endometrial distance association with expulsion risk | at 6 weeks after IUD placement
IUD-endometrial distance association with expulsion risk | at 3 months after IUD placement
IUD-endometrial distance association with expulsion risk | at 1 year after IUD placement

SECONDARY OUTCOMES:
Expected normal appearance of IUD on ultrasound and change in appearance over time | 6 weeks after IUD placement
Expected normal appearance of IUD on ultrasound and change in appearance over time | 3 months after IUD placement
Expected normal appearance of IUD on ultrasound and change in appearance over time | 1 year after IUD placement
IUD endometrial distance association with side effects | 6 weeks after IUD placement
IUD endometrial distance association with side effects | 1 year after IUD placement

CONTACTS AND LOCATIONS:
Overall Officials: Britt Lunde, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Elmhurst Hospital Center, Elmhurst, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Background] ACOG Practice Bulletin No. 121: Long-acting reversible contraception: Implants and intrauterine devices. Obstet Gynecol. 2011 Jul;118(1):184-196. doi: 10.1097/AOG.0b013e318227f05e. No abstract available. PMID 21691183
- [Background] Medical Eligibility Criteria for Contraceptive Use: A WHO Family Planning Cornerstone. 4th edition. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138639/ PMID 23741782
- [Background] Centers for Disease Control and Prevention (CDC). Update to CDC's U.S. Medical Eligibility Criteria for Contraceptive Use, 2010: revised recommendations for the use of hormonal contraception among women at high risk for HIV infection or infected with HIV. MMWR Morb Mortal Wkly Rep. 2012 Jun 22;61(24):449-52. PMID 22717514
- [Background] Levi E, Cantillo E, Ades V, Banks E, Murthy A. Immediate postplacental IUD insertion at cesarean delivery: a prospective cohort study. Contraception. 2012 Aug;86(2):102-5. doi: 10.1016/j.contraception.2011.11.019. Epub 2012 Jan 20. PMID 22264666
- [Background] Faundes D, Bahamondes L, Faundes A, Petta C, Diaz J, Marchi N. No relationship between the IUD position evaluated by ultrasound and complaints of bleeding and pain. Contraception. 1997 Jul;56(1):43-7. doi: 10.1016/s0010-7824(97)00072-3. PMID 9306030
- [Background] Faundes D, Perdigao A, Faundes A, Bahamondes L, Petta CA. T-shaped IUDs accommodate in their position during the first 3 months after insertion. Contraception. 2000 Oct;62(4):165-8. doi: 10.1016/s0010-7824(00)00167-0. PMID 11137069
- [Background] Shimoni N, Davis A, Westhoff C. Can ultrasound predict copper IUD expulsion after medical abortion? Poster presentation at NAF 2012 conference, Columbia University Medical Center.